CLINICAL TRIAL: NCT03859687
Title: A Randomized Controlled Trial of Antibody Responses by Vitamin Supplementation at the Time of Pneumococcus Vaccination in Children
Brief Title: Trial of Antibody Responses by Vitamin Supplementation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in starting recruitment
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCVIT
Record Dates: First submitted 2019-02-22; First posted 2019-03-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Children; Vitamin Supplements; PCV13; Hepatitis A vaccine
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): PCV (Prevnar-13 Vaccine) and the hepatitis A vaccine (Havrix Vaccine) plus a liquid oral vitamin A supplementation
  Interventions: Biological: Vitamin A supplementation
- Control group (Experimental): PCV (Prevnar-13 Vaccine) and the hepatitis A vaccine (Havrix Vaccine) only, 'No vitamin A supplementation'
  Interventions: Biological: No vitamin A supplementation

INTERVENTIONS:
Biological: Vitamin A supplementation — liquid oral vitamin A supplementation
  Arms: Intervention group
Biological: No vitamin A supplementation — No vitamin A supplementation
  Arms: Control group

SUMMARY:
Streptococcus pneumoniae, commonly called pneumococcus, can cause a wide range of diseases in children from mild ear infections to deadly pneumonia or meningitis. Vaccination is currently the single best way to protect children. Nutrition, especially the amount of vitamin A, may play a role in how well your body responds to infection or a vaccine. We call this an immune response. This research will look to see if children who take a vitamin with their vaccine have a better immune response than children who do not take a vitamin with their vaccine.

Primary Objective

To evaluate the influence of vitamin A supplementation on Prevnar vaccine immunogenicity based on changes in antibody scores in a commercial ELISA at Day 21 (after a booster vaccine dose) compared to pre-vaccine values.

Secondary Objectives

* To evaluate the relationship between baseline vitamin levels and pneumococcal or hepatitis A vaccine antibody responses (based on in commercial ELISAs) at Days 0 and 21.
* To evaluate the influence of vitamin A supplementation on hepatitis vaccine immunogenicity based on changes in antibody scores in a commercial ELISA at Day 21 compared to pre-vaccine values.
* To evaluate relationships between total serum antibodies (based on individual IgM, IgG1, IgG2, IgG3, IgG4, and IgA scores in a Luminex assay) at Day 0 and changes between Days 0 and 21 with baseline (Day 0) vitamin levels in young children, and with vitamin A supplementation.

DETAILED DESCRIPTION:
Children between the ages of 1 and 4 years old (inclusive) will be enrolled. All will receive PCV and hepatitis A vaccination. Those randomized to the treatment arm will receive 10,000 IU orally at the time of vaccination, while those randomized to the control arm will only receive vaccines. Vitamin levels and antibody responses towards the vaccines will be measured at screening, Day 0 (vaccination day) and Day +21. Children will be randomized using a stratified permuted block method.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 and 4 years old (inclusive) at the time of enrollment
* Fully weaned from breast-feeding or formula-feeding for at least 4 weeks prior to vaccination date (Day 0).
* Received at least 2 doses of Prevnar-13 vaccination
* Parent or legal guardian willing and able to provide informed consent.

Exclusion Criteria:

* Current use of investigational or immunosuppressive drugs (e.g., steroids) at the time of enrollment
* Parent/guardian planning to continue (or initiate) the administration of daily vitamin A, vitamin D, or multivitamin to the child during the study period.
* Evidence of developmental delay or evolving neurological disorders at screening.
* Current use of antibiotics or antivirals at enrollment.
* Currently receiving cancer related treatment.
* History of heart, kidney, or chronic respiratory condition (e.g., asthma) conditions.
* History of diabetes.
* Acute febrile illness [e.g., >100.0F (37.8oC) oral] illness within 3 days prior to enrollment.
* Received a previous PCV13 vaccine within 2 months of the enrollment date (Day 0).
* Received hepatitis A vaccine previously.
* Ever had a life-threatening allergic reaction to a dose of PCV13 vaccine, to an earlier pneumococcal vaccine called PCV7, or to any vaccine containing diptheria toxoid (for example, DTaP).

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate in two arms | Measured at Day 21
  The seroconversion rate, defined as the proportion of 4X increases or conversion from undetectable to detectable response in vaccine-specific antibody after vaccinations (Day 21) versus the baseline (Day 0) antibody level in intervention and control groups will be estimated and 95% confidence interval will be described for both groups. The 95% confidence interval will serve as a measure of precision of the seroconversion rate estimate. Chi-square test will be performed to make the comparison between two arms.
Sera titer ratio | Measured at Day 21
  Titer ratios will be summarized with descriptive statistics. Two-sample tests (t-test or Wilcoxon rank-sum test) will be applied whenever appropriate

SECONDARY OUTCOMES:
Spearman's correlation coefficient of vaccine antibody responses at days 0 with baseline vitamin levels for each arm. | Measured at Day 21
  Spearman's correlation coefficient.
Spearman's correlation coefficient of vaccine antibody responses at days 21 with baseline vitamin levels for each arm. | Measured at Day 21
  Spearman's correlation coefficient.
Proportion of subjects showing 4X increases or conversion from undetectable to detectable response in B cell responses after vaccinations for both groups, and by VA/VD stratum. | Measured at Day 21
  The proportion difference with 95% confidence interval will be reported via Chi-square test or Fisher's test.
Correlation of immunoglobulin M (IgM) antibody (measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 1 (IgG1) antibody (measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 2 (IgG2) antibody (measured by Luminex assay | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 3 (IgG3) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 4 (IgG4)antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin A (IgA) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient
Correlation of immunoglobulin M (IgM) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 2 (IgG2) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 3 (IgG3) antibody (measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin G subclass 4 (IgG4) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.
Correlation of immunoglobulin A (IgA) antibody(measured by Luminex assay) | Measured at Day 21
  Correlation will be expressed as Spearman's correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Nehali Patel, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org